CLINICAL TRIAL: NCT00350818
Title: Azacitidine Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for AML and MDS
Brief Title: Azacitidine Maintenance Therapy After Allogeneic Bone Marrow Transplantation (Allo BMT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0417
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Myelodysplastic Syndrome; Leukemia
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Allogeneic Transplantation; Leukemia; Azacitidine; Vidaza
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine (Experimental): Azacitidine after Allogeneic Transplantation
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — 8 mg/m^2 Subcutaneously Once Daily for 5 Days
  Other Names: Vidaza

SUMMARY:
Primary Objective:

-To determine the dose and schedule combination of 5-Azacitidine, when used as maintenance treatment after allogeneic transplantation for high-risk AML / MDS.

Secondary Objective:

-To assess the effect of treatment on survival after allogeneic transplantation for high-risk AML / MDS.

DETAILED DESCRIPTION:
Azacitidine is a drug that is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete medical history and physical exam. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will be given chemotherapy, before the transplant of donor cells. There are 2 major goals to giving this chemotherapy. One goal is to directly kill leukemic cells. The other goal is to block your ability to reject the donor cells that will be given to your for the transplantation.

All participants will receive a combination of 3 chemotherapy drugs--gemtuzumab, fludarabine, and melphalan. In order to receive gemtuzumab, your bone marrow leukemia cells have to be positive for a marker called "CD33," which is present in the majority of myeloid leukemias. If your cells are negative for that marker, the chemotherapy you receive will not include gemtuzumab. Anti-thymocyte globulin (ATG) will be given to patients receiving stem cells from an unrelated donor, or from a relative that is not fully matched with you.

All chemotherapy drugs are given by vein through a silicone catheter. Gemtuzumab is given 12 days before the transplant (may be given as an outpatient infusion). Fludarabine is given once a day for 4 days (5-2 days before the transplant), and melphalan is given as a single dose 2 days before the transplant. If you are receiving ATG, this drug will be given in 3 doses, given 3-1days before the transplant. The transplant day is usually referred to as "Day 0."

A total of 5 bone marrow biopsies will be collected during the first year after transplantation--before the start of treatment, around 1 month after transplantation, and around 4, 9, and 12 months after transplantation. To collect a bone marrow sample, an area of the hip bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. The bone marrow samples will be used primarily for disease status evaluation, but researchers will also use the samples for research on the way azacitidine works.

Eleven (11) blood samples (2 teaspoons each) will be collected for research purposes during the 1 year of your participation in this study. Samples will be collected before chemotherapy, before stem cell transplantation, before and after you receive 5-azacitidine (for each of the 4 cycles of treatment), and on the third week of the first cycle of 5-azacitidine treatment.

After the blood-forming cells are collected from the donor, they will be given to you by vein for your transplant. Before the infusion, you will receive medications, such as steroids and Benadryl (diphenhydramine), to decrease the risk of side effects. These "premedications" are given by vein usually 30 to 60 minutes before the transplant.

You will receive several medications to help the treatment work and to help decrease the risks of infections while your immune system is weak. Tacrolimus and methotrexate will be given to decrease the risk of graft-versus-host disease (GVHD), a problem that may occur if the donor's immune cells fight your body. Tacrolimus will be started 2 days before the transplant and will continue for a variable period of time (e.g., 3-12 months, or longer if you develop GVHD). Tacrolimus is given by vein at first and then by mouth, when patients are able to eat. Methotrexate is given by vein 1, 3, and 6 days after transplantation.

Several medications are used for the prevention of infections (potentially caused by fungal, bacterial, and viral organisms). Some of these antibiotics are given by vein, and some are given as pills, for variable lengths of time. You will receive medications while you are on tacrolimus or other medications that may weaken your immune system (such as steroids), in order to prevent infections, such as pneumonia. These antibiotics may include Bactrim, Diflucan, or other medications, if necessary.

You will be in the hospital for about 3-4 weeks after the transplant. You will have check-ups every day until you leave the hospital. After you leave, the frequency of clinic visits will vary, depending on your condition. You may need to come to the hospital as often as daily.

If your first bone marrow examination after transplantation determines that you are in remission, you will be eligible to receive azacitidine in one of 3 doses. Your dose and schedule of administration will be decided before you start the treatment. Participants will be enrolled starting with the smallest dose and moving upwards in terms of dose, if no side effects are detected. Each participant will have an assigned dose. This dose may be decreased or may be stopped or may not be given at all if certain side effects develop.

Azacitidine will be given as an injection under the skin once a day over 5 days in a row. This may be repeated once a month for up to 4 months after the transplant. You will be assigned to receive the drug for one to four cycles. You will have about 25 days of "rest" between each cycle of treatment (a cycle is the period of 1 month.). If intolerable side effects occur, treatment with azacitidine may be interrupted or stopped altogether before you finish treatment.

While on study, you will need to stay in Houston for up to 5 months after your transplant. You will then be required to return at 9 and 12 months after the transplant, though the frequency of the visits may be higher, if thought necessary by your doctor. After 1 year, your follow-up will continue as is standard of care for your disease.

This is an investigational study. Azacitidine and the other drugs described here are approved by the FDA. The use of azacitidine after allogeneic transplantation is experimental.About 90 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of AML (WHO classification: >=20% blasts in the bone marrow and / or peripheral blood), or MDS (IPSS intermediate-2 or higher) that at the time of allogeneic transplantation were in.
2. Induction Failure, relapsed disease or second or greater remission.
3. Patients in first complete remission that required more than 2 cycles of treatment to achieve the remission.
4. Donor: HLA-compatible related (HLA-A, -B, -DRB1 matched or with one-antigen mismatch) or
5. HLA-compatible unrelated (HLA-A, -B, -C and -DRB1 matched or with one-antigen mismatch)
6. Age 18 to 75 years and
7. Left ventricular ejection fraction >40% and
8. FEV1, FVC and DLCO >40% and
9. Serum creatinine <1.6 mg/dL and
10. Serum bilirubin < 1.6 mg/dL and
11. SGPT < 3 X upper limit of normal and
12. All patients and donors or guardian should be able to understand and sign informed consent.
13. Women of childbearing potential (any female who has experienced menarche, and who has not undergone surgical sterilization or is not post-menopausal) must have a negative serum pregnancy test.

Exclusion Criteria:

1. HIV positive
2. AML or MDS in first complete remission (defined as: bone marrow with less than 6% blasts, no circulating blasts, and a platelet count greater than 100,000 /mm^3.)
3. Active uncontrolled infection
4. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time to Toxicity | Baseline with 30 day cycles (up to 4 cycles), approximately 116 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcos de Lima, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org